CLINICAL TRIAL: NCT06650488
Title: Clopidogrel vs. Aspirin as Anti-thrombotic Therapy in Patients With S. Aureus Bacteremia
Acronym: Clopido-SNAP 2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Todd C. Lee MD MPH FIDSA (Other)
Responsible Party: Sponsor-Investigator, Todd C. Lee MD MPH FIDSA, Associate Professor of Medicine and Staff Scientist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-10899; 500048 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Staphylococcus Aureus Endocarditis; Staphylococcus Aureus Septicemia; Staphylococcus Aureus Bloodstream Infection
Keywords: S. aureus bactremia; S. aureus bloodstream infection; S. aureus endocarditis; aspirin; clopidogrel
MeSH Terms: interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Change to clopidogrel (Experimental): Patients will have their aspirin discontinued and start clopidogrel.
  Interventions: Drug: Clopidogrel
- Continue aspirin (Active Comparator): Patients will continue their existing aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — Patients will change from aspirin to clopidogrel (without loading dose)
  Arms: Change to clopidogrel
Drug: Aspirin — Patients will continue their existing aspirin.
  Arms: Continue aspirin

SUMMARY:
This is an open-label randomized controlled trial which will enroll patients with S. aureus bacteremia who are already taking aspirin for secondary prevention of cardiovascular events. We will randomize patients to continue their aspirin or change clopidogrel which is also approved for secondary prevention.

Unlike aspirin, clopidogrel may have activity against S. aureus. We wish to determine if changing to clopidogrel will improve outcomes in S. aureus bacteremia in people who otherwise would have a reason to be taking it.

This study is an approved sub-study of The Staphylococcus aureus Network Adaptive Platform (SNAP) trial (NCT05137119).

If positive, this study will support a Phase 3 RCT in people who do not currently have an indication for clopidogrel.

ELIGIBILITY:
The participant must meet all inclusion and exclusion criteria for the SNAP

Platform (NCT05137119) and also the following inclusion and exclusion criteria:

Inclusion Criteria:

* Patient is taking aspirin for secondary prevention of cardiovascular disease (coronary, cerebrovascular, or peripheral vascular disease)

Exclusion Criteria:

* Active bleeding (allowing up to 3 days from platform entry to randomize in the event anti-thrombotic therapy is resumed)
* Anticipated major cardiac surgery, neurosurgery, or spine surgery within the next 3 days
* Pregnancy
* Known receipt of clopidogrel, prasugrel, or ticagrelor within the last month
* Allergy to clopidogrel
* Concomitant receipt of oral Xa inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Desirability of Outcome Ranking (DOOR) | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Desirability of Outcome Ranking (DOOR) - an ordinal outcome with 5 levels defined:
  Rank 1 - Alive without complication Rank 2 - Alive with 1 complication Rank 3 - Alive with 2 complications Rank 4 - Alive with 3 complications Rank 5 - Dead
  Complications include:
  1. Clinical failure: Absence of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated.
  2. Infectious Complications: Including new endocarditis; new evidence of other deep metastatic foci (e.g., osteomyelitis or deep abscess); relapse of MRSA bacteremia after a patient has sterilized their initial blood cultures; readmission for subsequent care of S. aureus bacteremia; need for unplanned source control procedures
  3. Serious adverse drug event (Common Terminology Criteria class 4) due to study drug OR adverse drug event (classes 1-3) leading to discontinuation of the study drug

SECONDARY OUTCOMES:
Clinical Failure | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as the absence of resolution of clinical signs and symptoms of S. aureus bacteremia such that no additional antibiotic therapy is required or anticipated for its treatment.
Serious Adverse Event or Adverse Event Leading to Discontinuation | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as a serious adverse drug event (Common Terminology Criteria for Adverse Events (CTCAE) class 4) presumed due to study drug OR adverse drug event (CTCAE classes 1-3) leading to discontinuation of the study drug
All cause mortality | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Death from any cause
Infectious Complications | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Defined as change in therapy for inadequate clinical response; new endocarditis; new evidence of other deep metastatic foci (e.g., osteomyelitis or deep abscess); relapse of MRSA bacteremia after a patient has sterilized their initial blood cultures; readmission for subsequent care of S. aureus bacteremia; need for unplanned source control procedures. New implies that the complication was not suspected at enrollment and is not a function of delay to diagnostic testing.
Clinically relevant major bleeding | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  This will be defined according to the criteria of the International Society on Thrombosis and Haemostasis as one or more of the following: fatal bleeding; symptomatic bleeding in a critical area or organ (including hemorrhagic stroke); bleeding that causes a fall in hemoglobin level of ≥20 g/L; or bleeding that requires a transfusion of 2 or more units of whole blood or red cells. For bleeds into non-critical areas, we will also record the site of bleeding.
Clinically relevant venous thromboembolic events | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  This will be defined as an acute objectively confirmed deep vein thrombosis (upper extremity, lower extremity, other such as portal vein, cerebral vein, splanchnic vein) and/or segment or proximal pulmonary embolism, which is symptomatic and/or necessitates specific treatment. Below knee DVT and superficial thrombophlebitis are not included. Pulmonary embolism needs to be, segmental or proximal. Subsegmental pulmonary embolisms are not included as they have poor interrater reliability and may represent artefact in up to 50% of cases.
Clinically relevant stroke | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Stroke is defined as the acute onset of focal neurological dysfunction caused by brain, spinal cord, or retinal vascular injury because of infarction (ischemia). Ideally, at least one of the following should be present to confirm the diagnosis of stroke: confirmation by neurology, stroke specialist, or neurosurgical specialist, brain imaging (e.g., CT scan, MRI scan, or cerebral vessel angiography compatible with acute ischemia). If the acute focal signs represent a worsening of a previous deficit, these signs must persist for more than 24 hours and be accompanied by an appropriate new MRI or CT scan finding. In the absence of neuroimaging, a staff neurologist consult which makes the diagnosis of stroke will be considered.
Clinically relevant acute myocardial infarction | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Patients with S. aureus bacteremia often have substantial physiological stresses which can be associated with rises in cardiac troponin (demand ischemia). For the purposes of this outcome, acute myocardial infarction is captured as a type 1 myocardial infarction: detection of rise and/or fall of cardiac biomarkers with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia. For the purposes of this pragmatic trial, such a myocardial infarction will be inferred from the opinions of the staff cardiologist, intensivist, or general internal medicine specialist. The peak troponin value will be recorded, and a redacted copy of the relevant consultant's note and ECGs will be uploaded for audit.
Clinically relevant arterial thromboembolic event | Day 90 post enrollment in the S. aureus Network Adaptive Platform Trial (NCT05137119)
  Clinical history compatible with sudden worsening of end organ or limb perfusion and confirmation by imaging (e.g., CT angiography, arterial doppler) or need for urgent surgery or thrombolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD MPH FIDSA, Principal Investigator — Research Institute of the McGill University Health Centre; Emily G McDonald, MD MSc, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre (Royal Victoria Hospital and Montreal General Hospital), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing policies are dependent on the policies of the SNAP Platform (NCT05137119)

REFERENCES:
- [Background] Gentry CA, Williams RJ 2nd, Whitman CM, Thind SK, Kliewer BS. Staphylococcus aureus bacteraemia treatment outcomes in patients receiving ticagrelor vs a propensity-matched cohort receiving clopidogrel. Int J Antimicrob Agents. 2023 Apr;61(4):106743. doi: 10.1016/j.ijantimicag.2023.106743. Epub 2023 Feb 2. PMID 36736927
- [Background] Tong SYC, Mora J, Bowen AC, Cheng MP, Daneman N, Goodman AL, Heriot GS, Lee TC, Lewis RJ, Lye DC, Mahar RK, Marsh J, McGlothlin A, McQuilten Z, Morpeth SC, Paterson DL, Price DJ, Roberts JA, Robinson JO, van Hal SJ, Walls G, Webb SA, Whiteway L, Yahav D, Davis JS; Staphylococcus aureus Network Adaptive Platform (SNAP) Study Group. The Staphylococcus aureus Network Adaptive Platform Trial Protocol: New Tools for an Old Foe. Clin Infect Dis. 2022 Nov 30;75(11):2027-2034. doi: 10.1093/cid/ciac476. PMID 35717634
- [Background] Caffrey AR, Appaneal HJ, LaPlante KL, Lopes VV, Ulloa ER, Nizet V, Sakoulas G. Impact of Clopidogrel on Clinical Outcomes in Patients with Staphylococcus aureus Bacteremia: a National Retrospective Cohort Study. Antimicrob Agents Chemother. 2022 Jun 21;66(6):e0211721. doi: 10.1128/aac.02117-21. Epub 2022 Apr 13. PMID 35416712
- See also: Main Website for the S. aureus Network Adaptive Platform Trial (SNAP) — https://www.snaptrial.com.au/